CLINICAL TRIAL: NCT04632433
Title: A Phase II, Single Arm Study Investigating Neoadjuvant Plus Adjuvant Treatment With Cemiplimab in High Risk, Surgically Resectable, Stage III Cutaneaous Squamous Cell Carcinoma
Brief Title: Neoadjuvant Plus Adjuvant Treatment With Cemiplimab in Cutaneaous Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Melanoma Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO-CESQ
Record Dates: First submitted 2020-11-06; First posted 2020-11-17 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cutaneous Squamous Cell Carcinoma
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Intervention Model Description: Patients will receive cemiplimab at a dosage of 350 mg every 3 weeks for two cycles prior surgery. Stage III stage must be documented at screening and re-assessed prior surgery by spiral or multidetector computed tomography (CT) scan (if clinically indicated) and Positron emission tomography (PET). Postoperatively, adjuvant immunotherapy with cemiplimab will be administered at a dosage of 350 mg every 3 weeks for one year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental): Patients will receive cemiplimab at a dosage of 350 mg every 3 weeks for two cycles prior surgery. Stage III stage must be documented at screening and re-assessed prior surgery by spiral or multidetector computed tomography (CT) scan (if clinically indicated) and Positron emission tomography (PET). Postoperatively, adjuvant immunotherapy with cemiplimab will be administered at a dosage of 350 mg every 3 weeks for one year.
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — 350 mg every 3 weeks

SUMMARY:
Neoadjuvant plus adjuvant treatment with immunotherapy may have an anti-tumor activity and reduce the risk of relapse in patients with high risk surgically resectable stage III cutaneous squamous cell carcinoma.

DETAILED DESCRIPTION:
Cutaneous squamous cell carcinoma (CSCC) is the second most common skin cancer in US. It is associated with a surgical cure rate >95% in early stage disease but a small percentage of patients develop unresectable locally advanced or metastatic CSCC. The 2018 FDA approval of Libtayo was based on a combined analysis of data from an open-label, multi-center, non-randomized Phase 2 trial known as EMPOWER-CSCC-1 (Study 1540) and two advanced CSCC expansion cohorts from a multi-center, open-label, non-randomized Phase 1 trial (Study 1423). Conventional cytotoxic chemotherapy can induce tumor responses but is often poorly tolerated, specially among older patients with CSCC. CSCC has higher mutation burden than any tumor type and immunosuppression is a known risk factor. Furthermore, PD-L1 expression has been associated with high risk disease1 suggesting that CSCC may be responsive to PD-1 checkpoint blockade.

Cemiplimab is a human anti-PD-1 monoclonal antibody, under study for patients with unresectable locally advanced and/or regionally or metastatic CSCC. It has been studied in a phase I dose escalation, where a durable radiologic complete response was achieved in CSCC patients.2-3 In this study, the partial response was 25% in locally advanced and 60% in metastatic CSCC,stable disease was 31.3% in locally advanced and 10% in metastatic CSCC, progressive disease was 25% in locally advanced and 20% in metastatic CSCC with an overall response rate of 46.2% and a disease control rate of 69.2%. The 2018 FDA approval of Libtayo was based on a combined analysis of data from an open-label, multi-center, non-randomized Phase 2 trial known as EMPOWER-CSCC-1 (Study 1540) and two advanced CSCC expansion cohorts from a multi-center, open-label, non-randomized Phase 1 trial (Study 1423). Together, the trials represent the largest prospective data set in advanced CSCC. The major efficacy outcome measures for the integrated analysis of EMPOWER-CSCC-1 and the two CSCC expansion cohorts were confirmed objective response rate (ORR), as assessed by independent central review (ICR), and ICR-assessed duration of response (DOR).

Across the entire population, the overall response rate (ORR) at a median follow-up of 8.9 months was 47% (95% CI, 38-47). The complete response (CR) rate was 4% and the partial response (PR) rate was 44%. The duration of response ranged from 1 month to over 15 months. Sixty-one percent of patients had a duration of response ≥6 months.

Among 75 patients with metastatic CSCC, the ORR was 47% (95% CI, 35-59). The CR rate was 5% and the PR rate was 41%. The duration of response ranged from 3 months to over 15 months. Sixty percent of patients had a duration of response ≥6 months. In the 33 patients with locally advanced disease, the ORR was 49% (95% CI, 31-67), comprising all PRs. The duration of response ranged from 1 month to over 13 months. Sixty-three percent of patients had a duration of response ≥6 months.

Cemiplimab therefore produced rapid, deep and durable tumor reductions in target lesions.

Cemiplimab appears to be active regardless PD-L1 expressione in the tumor and no apparent association between PD-L1 IHC results and objective responses was determined. Cemiplimab was generally well tolerated in CSCC, and most commonly associated with fatigue (23.1% prevalence), arthralgia, rash maculopapular, diarrhea, nausea, hypothyroidism (7.7%) of any grade.

The advantage of neoadjuvant trials is the availability of blood and tumor tissue samples before and after systemic therapy for the conduct of novel mechanistic and biomarker studies in the circulation and the tumor microenvironment.

Based on the available results to date, the investigators aim to conduct a phase II single arm trial to define the role of neoadjuvant plus adjuvant immunotherapy in patients with stage III CSCC. This approach has the potential to define whether neoadjuvant treatment with cemiplimab has antitumor activity and whether it reduces the risk of relapse after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged ≥18 years.
2. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
3. Patients must have histologically or cytologically confrimed stage III cutaneous squamous cell carcinomas. The definition of resectability can be determined by the patient's surgical oncologist and verified via discussion at Multidisciplinary Tumor Conference attended by CSCC medical and surgical oncology staff. Resectable tumors are defined as having no significant vascular, neural or bony involvement.
4. Patients must be medically fit enough to undergo surgery as determined by the surgical oncology team.
5. Patients must have measurable disease, defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
7. Patients must have organ and marrow function
8. Female subjects of childbearing potential must have a negative pregnancy test result at baseline and must practice a reliable method of contraception for the total study duration plus 16 weeks (i.e., 30 days plus the time required for cemiplimab to undergo five half lives) after the last dose of cemiplimab.
9. Men who are sexually active with women of childbearing potential must practice a reliable method of contraception for the total study duration plus 16 weeks (i.e., 80 days plus the time required for cemiplimab to undergo five half-lives) after the last dose of cemiplimab.

Exclusion Criteria:

1. Evidence of metastatic disease extra lymphnodal.
2. Currently and previous cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug.
3. Prior malignancy within the prior 5 years, except for the following: in-situ cervical cancer, thyroid cancer (except anaplastic) or any cancer from which the patient has been disease-free for 2 years.
4. Any major surgery within the last 3 weeks.
5. Unwillingness or inability to follow the procedures required in the protocol.
6. Uncontrolled diabetes, hypertension, pneumonitis and abnormal thyroid function or other medical conditions that may interfere with assessment of toxicity.
7. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of treatment.
8. Female subjects who are pregnant (positive pregnancy test), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
9. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection;
10. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate | 43-71 days
  <10% remaining viable tumour cells in resected primary tumor

SECONDARY OUTCOMES:
Recurrence-free survival | At 6 and 12 months postoperative
  RFS - the time from start of treatment until disease recurrence (local, regional or distant) or death from any cause
Overall Survival | Until three years from last infusion
  OS - the time from the date of first dose until the date of death from any cause
Prevalence of related AEs | Through study treatment completion, an average of 17 months
  Number of participants with treatment-related adverse events by grade as assessed by CTCAE v5.0
Use of selected biomarkers to detect molecular and immunophenotypic changes | At screening 1 and 2, at surgery, every 12 weeks during adjuvant and at recurrence of disease untill an average of 1 year from surgery
  Predictive biomarkers and thier changes in tumor and blood samples will be correlated with pathological response and patient's outcome

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Ascierto, MD, Study Chair — Fondazione Melanoma Onlus
Locations (7):
- Italy (7):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, Bergamo
  - Ospedale S.M. Annunziata - Azienda USL Toscana Centro, Bagno a Ripoli, Firenze
  - IRCCS - Istituto Scientifico Romagnolo per la Cura e lo Studio dei Tumori (I.R.S.T) S.r.l., Meldola, Forlì-Cesena
  - Fondazione I.R.C.C.S. Istituto Nazionale dei Tumori, Milan, Milano
  - Istituto Nazionale per lo Studio e la Cura dei Tumori "Fondazione Giovanni Pascale", Naples, Naples
  - Istituto Oncologico Veneto, Padua, Padova
  - ASST Spedali Civili Brescia, Brescia

IPD SHARING:
Plan to Share IPD: No